CLINICAL TRIAL: NCT05773703
Title: A Phase 0 Study of the Pharmacokinetics and Biodistribution of PSMA-Targeted [In-111]-Labeled Trillium Compounds With and Without PTI-122 in Patients With Metastatic Prostate Cancer to Inform Future Phase 1 Dosing With [Ac-225]-Trillium-PSMA Radionuclide Therapy
Brief Title: Exploratory PK and Imaging Study of PSMA-Targeted Trillium Compounds and PTI-122 in Metastatic Prostate Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Ratio Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: RTX-PSMA-P101
Record Dates: First submitted 2023-02-23; First posted 2023-03-17 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Each Trillium Compound will first be evaluated alone, then with single doses (5, 10, 15 mg) of the cytoprotective agent, PTI-122. Trillium Compound with two doses of PTI-122 at the preferred dose level may be studied if indicated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Trillium Compound Alone (Experimental): Single dose of PSMA-Targeted [In-111]-Labeled Trillium Compound
  Interventions: Drug: PSMA-Targeted [In-111]-Labeled Trillium Compound
- Trillium Compound + Single Dose PTI-122 (Experimental): Single dose of PSMA-Targeted [In-111]-Labeled Trillium Compound plus single dose of PTI-122 at 5, 10 or 15 mg
  Interventions: Drug: PSMA-Targeted [In-111]-Labeled Trillium Compound; Drug: PTI-122
- Trillium Compound + Multiple Dose PTI-122 (Experimental): Single dose of PSMA-Targeted [In-111]-Labeled Trillium Compound plus two doses of PTI-122 at the preferred dose level
  Interventions: Drug: PSMA-Targeted [In-111]-Labeled Trillium Compound; Drug: PTI-122

INTERVENTIONS:
Drug: PSMA-Targeted [In-111]-Labeled Trillium Compound — Radiotracer
Drug: PTI-122 — Cytoprotective agent
  Arms: Trillium Compound + Multiple Dose PTI-122; Trillium Compound + Single Dose PTI-122

SUMMARY:
Exploratory study in adult males with metastatic prostate cancer intended to characterize the pharmacokinetics and biodistribution of PSMA-Targeted [In-111]-Labeled Trillium Compounds with and without the cytoprotective agent PTI-122. Up to 36 eligible subjects will be enrolled. Additional subjects may be enrolled if there is insufficient data for evaluation, for example if the original study subjects do not complete required imaging studies for reasons unrelated to adverse events.

Up to four PSMA-Targeted [In-111]-Labeled Trillium Compounds will be evaluated. Each compound will be evaluated first without the cytoprotective agent, PTI-122, then the [In-111]-labeled Trillium Compound may be co-administered with PTI-122.

ELIGIBILITY:
Inclusion Criteria:

* Adult males with metastatic prostate cancer
* ECOG performance score 0-2
* Stable androgen deprivation or other hormone therapy (30 days) or therapy planned but not yet initiated
* PSMA PET scan between 3 and 28 days prior to radiotracer injection with at least 2 PSMA positive lesions and either:

  1. One soft tissue lesion measuring ≥ 15 mm in the longest diameter with SUVmax lesion ≥ SUVmean normal liver, OR
  2. Two bone lesions measuring ≥ 15 mm in the longest diameter with SUVmax lesion ≥ 2 x SUVmax normal liver
* Able to understand and adhere to study requirements, and voluntarily give informed consent

Exclusion Criteria:

* No other malignancy undergoing treatment
* No PSMA-targeted therapy ongoing
* Inability or unwillingness to undergo SPECT/CT imaging
* Serum creatinine > 1.5 mg/dL or creatinine clearance ≤50 mL/min by Cockcroft-Gault estimation
* Concurrent participation in the active treatment phase of another clinical trial of investigational medicinal product(s)
* Significant intercurrent illness, treatment-related toxicity, or psychiatric illness/social situation that could place the subject at undue risk during study participation, significantly alter study outcomes, or affect subject compliance with study requirements for dosing and evaluation, as determined by the investigator

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Males with prostate cancer
Enrollment: 23 (Actual)
Dates: Start 2022-12-08 (Actual); Primary Completion 2023-12-12 (Actual); Study Completion 2023-12-12 (Actual)

PRIMARY OUTCOMES:
Amount of radiotracer absorbed by tumor | Over 168 hours post-injection
  Tumor uptake measured on imaging
Amount of radioactivity in blood | Over 168 hours post-injection
  Radioactivity measured pre- and post-radiotracer injection
Amount of radiotracer absorbed by organs | Over 168 hours post-injection
  Organ uptake measured on imaging

SECONDARY OUTCOMES:
Amount of PTI-122 in blood | Over 168 hours post-injection
  PTI-122 measured pre- and post-dose
Incidence of adverse events | Over 168 hours post-injection
  Occurrence of adverse events during the study

CONTACTS AND LOCATIONS:
Overall Officials: John Babich, PhD, Study Director — Ratio Therapeutics, Inc.
Locations (4):
- United States (4):
  - Biogenix Molecular, Miami, Florida
  - Advanced Molecular Imaging & Therapy, Glen Burnie, Maryland
  - XCancer Omaha/Urology Cancer Center, Omaha, Nebraska
  - University of Tennessee Medical Center, Knoxville, Tennessee

IPD SHARING:
Plan to Share IPD: No